CLINICAL TRIAL: NCT03079193
Title: Post Thyroidectomy Endoscopic Laryngeal Examination :Is it Mandatory?
Status: Completed | Type: Observational
Sponsor: Khamis Mushayt General Hospital (Other Government)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, wagih ghnnam, associate professor of general surgery, Khamis Mushayt General Hospital
Other Study IDs: khamisMGH WA1
Record Dates: First submitted 2014-03-13; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Thyroid
Keywords: post thyroidectomy; laryngeoscopic examination
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- videoscopic laryngeal examination: 50 patients post thyroidectomy will do mandatory post thyroidectomy videoscopic examination of the larynx
- No vedioscopic larygeoscopic examination: 50 patients post thyroidectomy will be followed up and will not do vedeoscopic videoscopic laryngeal examination routinely they will do it if indicated

SUMMARY:
Post thyroidectomy laryngeal nerve injuries are frequently encountered specially in total and near total thyroidectomy some unilateral injuries are not clinically evident and asymptomatic.

The aim of this study is to compare mandatory versus selective post-thyroidectomy endoscopic examination of larynx to detect laryngeal nerve injuries.

DETAILED DESCRIPTION:
100 patients were randomly divided into two groups, group I for whom mandatory post thyroidectomy endoscopic laryngoscopic examination and the other group of only symptomatic patients selected for direct laryngoscopic examination.

ELIGIBILITY:
Inclusion Criteria:

* all post thyroidectomy patients

Exclusion Criteria:

-

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 patients post thyroidectomy will be randomly divided into two groups group I for whom mandatory vedioscopic laryngeal examination is done while the other group II patients for whom no routine vedioscopic laryngeal examination done only if symptoms developed
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
endoscopic laryngeal examination post thyroidectomy | 3 years
  usefulness of endoscopic laryngeal examination post thyroidectomy

IPD SHARING:
Plan to Share IPD: Undecided